CLINICAL TRIAL: NCT02367547
Title: Superficial Basal Cell Cancer's Photodynamic Therapy: Comparing Three Photosensitizers: Hexylaminolevulinate and Aminolevulinic Acid Nano Emulsion Versus Methylaminolevulinate
Brief Title: Superficial Basal Cell Cancer's Photodynamic Therapy: Comparing Three Photosensitizers: HAL and BF-200 ALA Versus MAL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Tampere University (Other); University of Jyvaskyla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JointAPHSHC; 2014-002746-50 (EudraCT Number)
Record Dates: First submitted 2015-01-31; First posted 2015-02-20 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Neoplasms, Basal Cell; Carcinoma, Basal Cell; Photochemotherapy; Photosensitizing Agents
MeSH Terms: conditions — Neoplasms, Basal Cell; Carcinoma, Basal Cell | interventions — 5-aminolevulinic acid hexyl ester; Aminolevulinic Acid; BF-200 ALA; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hexylaminolevulinate cream (Experimental): 2% Hexylaminolevulinate (Hexvix, Photocure) mixed with Unguentum M (Allmiral) cream
  Interventions: Drug: Hexylaminolevulinate cream
- Aminolevulinic Acid Nano Emulsion (Experimental): 78 mg/g Aminolevulinic Acid Nano Emulsion
  Interventions: Drug: Aminolevulinic Acid Nano Emulsion
- Methylaminolevulinate cream (Active Comparator): 160 mg/g Methylaminolevulinate cream
  Interventions: Drug: Methylaminolevulinate cream

INTERVENTIONS:
Drug: Hexylaminolevulinate cream — The cream is mixed up by the Pharmacy Yliopiston Apteekki for the study and every set is analysed by mass spectrometry.
  Other Names: HAL; Hexvix, Photocure
  Arms: Hexylaminolevulinate cream
Drug: Aminolevulinic Acid Nano Emulsion — In the study we use Ameluz.
  Other Names: Ameluz, Biofrontera; L01XD04; BF-200 ALA
  Arms: Aminolevulinic Acid Nano Emulsion
Drug: Methylaminolevulinate cream — In the study we use Metvix.
  Other Names: Metvix, Galderma; L01X D03; MAL
  Arms: Methylaminolevulinate cream

SUMMARY:
This pilot study compares three photosensitisers, hexylaminolevulinate (HAL) and aminolevulinic acid nano emulsion (BF-200 ALA) to methylaminolevulinate (MAL) in photodynamic therapy of superficially growing basal cell carcinomas. Study is conducted using randomised prospective double blinded comparing design. Fluorescence is measured in A.U. (Arbitrary Unit) with standardised set-up before and after the exposure. Efficacy is assessed clinically, histologically and by hyperspectral imaging system at 3 months, 12 months and 5 years.

DETAILED DESCRIPTION:
Study recruits volunteering patients, who are referred to the department of dermatology and allergology, Päijät-Häme Central Hospital, Lahti, with 99 clinically assessed superficial basal cell carcinoma on the body area, not face and scalp. Diagnoses is confirmed histologically by punch biopsies and hyperspectral images are taken before the biopsies. The lesions are randomised in three groups: interventions HAL and BF-200 ALA and comparator MAL. Photodynamic therapy is given by the standard procedure. Fluorescence is measured in A.U. (Arbitrary Unit) with standardised set-up, with Wood's light, digital camera and a yellow lens, before and after the exposure. Pain is measured in VAS-scale before, during and after the exposure. Efficacy is assessed clinically, histologically and by hyperspectral imaging system at 3 months, 12 months and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* superficial basal cell carcinomas on body area (clinically assessed to be mainly superficially growing and later on a biopsy proven sBCC or thin nBCC)
* lesions accepted needs to be 10 cm apart from each other

Exclusion Criteria:

* pigmented, morpheaform, infiltrative or nodular basal cell carcinomas
* lesions that are in face and scalp area
* pregnancy
* breast feeding
* allergy to photosensitizer
* phorphyria or photosensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Histological lesion clearance | 3 months
Histological lesion clearance | 12 months
Histological lesion clearance | 5 years

SECONDARY OUTCOMES:
Detection of subclinical lesion with hyperspectral imaging system | 3 months
Detection of subclinical lesion with hyperspectral imaging system | 12 months
Detection of subclinical lesion with hyperspectral imaging system | 5 years

OTHER OUTCOMES:
Fluorescence measured in A.U. (Arbitrary Units) with standardised set-up, with Wood's light, digital camera and a yellow lens | before (point 0 min) and after (point 8 min) the exposure
Pain in VAS-scale | in the beginning (point 0 min), middle (point 4 min) and end (point 8 min) of the exposure

CONTACTS AND LOCATIONS:
Overall Officials: Mari Grönroos, MD, PhD, Study Director — Päijänne Tavastia Central Hospital; Mari K Salmivuori, MD, Principal Investigator — Päijänne Tavastia Central Hospital
Locations (1):
- Joint Authority for Päijät-Häme Social and Health Care, Lahti, Finland